CLINICAL TRIAL: NCT06301828
Title: A Prospective, Single-arm Clinical Study of Endostar Combined With Stereotactic Body Radiation Therapy and Envafolimab in the Treatment of Advanced Gastrointestinal Tumors After Multi-line Treatment
Brief Title: Endostar Combined With SBRT and Envafolimab in the Treatment of Advanced Gastrointestinal Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY202401
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-02

CONDITIONS: Gastrointestinal Neoplasms
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — envafolimab; endostar protein; Endostatins

STUDY DESIGN:
Intervention Model Description: Gastrointestinal neoplasms
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Enrolled patients were treated with endostar combined with stereotactic body radiation therapy and Envafolimab.
  Interventions: Drug: Envafolimab Injection; Drug: Endostar

INTERVENTIONS:
Drug: Envafolimab Injection — Endostar+SBRT+Envafolimab Injection
  Other Names: KN035
Drug: Endostar — Endostar+SBRT+Envafolimab Injection
  Other Names: Recombinant Human Endostatin Injection

SUMMARY:
This is a single-arm, prospective, exploratory clinical study to evaluate the efficacy and safety of endostar combined with stereotactic body radiation therapy (SBRT) and Envafolimab in patients with advanced gastrointestinal cancer after multi-line treatment.

DETAILED DESCRIPTION:
This is a single-arm, prospective and exploratory clinical study. Sixteen patients with gastric or colorectal cancer who did not have standard treatment or refused standard treatment/chemotherapy after multi-line treatment were enrolled. The patients were treated with endostar combined with stereotactic body radiation therapy (SBRT) and Envafolimab to evaluate the efficacy and safety of this regimen. The primary endpoints were objective response rate (ORR) and disease control rate (DCR). The secondary endpoints were safety, progression-free survival (PFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years old, regardless of gender
* advanced gastrointestinal tumors confirmed by histopathology or cytology;
* patients with gastrointestinal tumors who did not or refused standard treatment at enrollment；Each line of treatment for advanced disease includes one or more drugs for one or more cycles； The pre-permissible treatment was combined with molecular targeted drugs (except endostar)； Patients with previous PD-1 treatment were eligible
* ECOG-PS score of 0-2
* The main organ function was normal and met the following requirements: Blood routine examination (no blood transfusion within 14 days) : a. HB≥80g/L; b. ANC ≥1.5×109/L; c. PLT ≥60×109/L; ② Biochemical examination should meet the following criteria: a. BIL<1.5 times the upper limit of normal (ULN); b. ALT and AST<2.5×ULN; ALT and AST< 5×ULN，if liver metastasis was present; c. Serum Cr≤1×ULN, endogenous creatinine clearance ≥50ml/min (Cockcroft-Gault formula)
* predicted survival time ≥3 months
* Patients voluntarily participated in this study and signed the informed consent form (ICF)

Exclusion Criteria:

* hypertensive patients whose blood pressure could not be reduced to normal range by antihypertensive drugs (systolic blood pressure>140 mmHg/diastolic blood pressure >90 mmHg); Patients with ≥ grade Ⅱ coronary artery disease, arrhythmia (including QTc prolongation > 450 ms in men and > 470 ms in women) and cardiac insufficiency
* patients with active immune diseases
* abnormal coagulation function (INR>1.5×ULN, APTT>1.5×ULN) with bleeding tendency
* symptomatic central nervous system metastasis
* pregnant or lactating women
* Other patients deemed ineligible for enrollment by the treating physician

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2025-06-21 (Estimated); Study Completion 2026-02-21 (Estimated)

PRIMARY OUTCOMES:
DCR | 12 months after the last subject participating in
  The proportion of subjects with complete response (CR), partial response (PR)and stable disease in(SD) in total subjects
ORR | 12 months after the last subject participating in
  The proportion of subjects with complete response (CR) and partial response (PR) in total subjects

SECONDARY OUTCOMES:
PFS | 12 months after the last subject participating in
  Progression-free survival (PFS per RECIST 1.1) is defined as the time from randomization to the date of first documentation of disease progression or death, whichever occurs first.
Incidence of Treatment-Emergent Adverse Events | Up to 2 years
  Occurrence and severity of AEs by NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: wei X wei, M.D., Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No